CLINICAL TRIAL: NCT04741035
Title: Effectiveness of Modified Sternal Precautions Versus Conventional Sternal Precautions in Improving Physical Function After Sternotomy
Brief Title: Modified Sternal Precautions Versus Conventional Sternal Precautions in Physical Function After Sternotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC00707 Huma Balqias
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases
Keywords: Sternal precautions; Sternal restrictions; CABG
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified sternal precautions (Experimental): Interventional group (Modified sternal precautions)
  Interventions: Other: Modified sternal precautions
- Conventional sternal precautions (Active Comparator): Control group (Conventional sternal precautions)
  Interventions: Other: Conventional sternal precautions

INTERVENTIONS:
Other: Modified sternal precautions — Use pain and discomfort to guide the safe use of the arms Avoid pushing or pulling with one arm Use both arms close to the body during lifting Use of arms is possible, but keep them close to the body Avoid stretching one or both arms backwards at the same time Use a cushion or perform sternal preservation technique (crossing the arms in a 'self-hugging 'posture) when coughing.
  When transferring, roll onto the side, ease the legs over the edge of the bed and carefully use the arms to sit up from a lying position
  Arms: Modified sternal precautions
Other: Conventional sternal precautions — Avoid pushing or pulling through the arms Avoid one-arm (unilateral) activity Limit the elevation of the arms to 90 degrees Avoid lifting objects heavier than 2 kg Use a cushion or perform sternal preservation technique (crossing the arms in a 'self-hugging' posture) when coughing Limit the use of the arms when transferring from sitting to standing and getting out of bed Avoid placing the arms behind the back
  Arms: Conventional sternal precautions

SUMMARY:
This research study Effectiveness of modified sternal precautions versus conventional sternal precautions in improving physical function after sternotomy .After recruitment of the subjects, the intervention group will receive modified sternal precaution while the control group will receive conventional sternal precautions and they will be assess for their physical activity, kinesiophobia, quality of life and post sternotomy pain.

DETAILED DESCRIPTION:
This study will address the scarcity of research and the variations in recommendations regarding sternal precautions and restrictions of upper limb movement in cardiac patients and will help to evaluate the effect of modified sternal precautions on patients' pain and functional activity. As physical therapists are the ones who have maximum exposure to practice and teaching of sternal precautions, therefore this study will help to formulate the guidelines regarding the use of upper limb during cardiac rehabilitation exercises and making standards for sternal precautions and its management following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Open heart surgery patients (CABG and Valve surgeries)

Exclusion Criteria:

* Unstable vitals
* Patient needing maximum assistance
* Decline consent

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 40 and above
Enrollment: 40 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Short physical performance battery | 4 Week
  SPBB is a commonly used tool in clinical setting for measuring the physical performance of patients. It is known for its feasibility and shorter time to conduct. It has been used in different studies for reporting outcome measure post cardiac surgery. This outcome measure is also selected due to its high validity and reliability. The reliability of the test is 0.87. It is divided into three subtests: balance, a short walk at normal pace and lastly standing up from a chair five times repeatedly. These subsets exemplify core tasks being important for independent living.
Functional difficulties questionnaire | 4 week
  Functional difficulties questionnaire is a functional outcome measures that specially focuses on the thoracic region and upper limb movements in people following cardiac surgery. The validity of the questionnaire is 0.971 while its reliability is 0.918. The questionnaire is divided into 13 questions which consists of functional tasks, causing difficulty following cardiac surgery. Participants are required to mark on an unmarked 10cm VAS the level of difficulty they experienced when completing each of the included tasks, based on the previous time they experience.
Tampa scale of Kinesiophobia (TSK-II) | 4 week
  It is a broadly used tool to measure pain related fear beliefs regarding movement and re-injury. The validly of the questionnaire range between 0.74 to 0.87 and its reliability is 0.747. It is a self-reported questionnaire. It includes 11 questions scale on likert scale ranging from 1 to 4 where 1 means strongly disagree while 4 means strongly agree. The total score ranges between 11 to 44. Higher score indicate high level of kinesiopobhia. A reduction of points equal or more than 3 points accounting for about 10% is considered as relevant change.
Mcgill pain questionnaire - short form version 2 (SF-MPQ-2) | 4 Week
  It is one of the most widely used questionnaire for the measurement of pain. Its benefit is that it provides valuable information on the sensory, affective and evaluative dimensions of pain experience by an individual. It has a capability of discriminating among different types of pain problems. It has become one of the most commonly used tests for the measurement of pain following cardiac surgery via sternotomy. The reliability of the questionnaire ranges from 0.75 to 0.83.

SECONDARY OUTCOMES:
Health survey (SF-36) | 4 week
  This questionnaire provides overall measure of quality of recovery of patient according to the patient's perspective. It is a reliable and valid tool used mainly in clinical practices to measure health related quality of life following cardiac surgery. The reliability of scale is 0.65 to 0.96. This tool consists of eight domains comprising of physical functioning, role physical functioning, role emotional functioning, mental health, vitality, social functioning, bodily pain and general health. Responses are recorded on a five-point Likert scale and then transformed onto a 100-point scale. Score higher than 50 shows better health state and less pain experienced

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid, MS, Principal Investigator — Riphah International University
Locations (1):
- Rehman medical institute, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein AJ, Polsky D, Yang F, Yang L, Groeneveld PW. Coronary revascularization trends in the United States, 2001-2008. JAMA. 2011 May 4;305(17):1769-76. doi: 10.1001/jama.2011.551. PMID 21540420
- [Background] Deb S, Wijeysundera HC, Ko DT, Tsubota H, Hill S, Fremes SE. Coronary artery bypass graft surgery vs percutaneous interventions in coronary revascularization: a systematic review. JAMA. 2013 Nov 20;310(19):2086-95. doi: 10.1001/jama.2013.281718. PMID 24240936
- [Background] Hodge T. Fast Facts for the Cardiac Surgery Nurse: Caring for Cardiac Surgery Patients in a Nutshell: Springer Publishing Company; 2015.
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):399-410. doi: 10.1161/01.cir.0000442015.53336.12. No abstract available. PMID 24446411
- [Background] Price KJ, Gordon BA, Bird SR, Benson AC. A review of guidelines for cardiac rehabilitation exercise programmes: Is there an international consensus? Eur J Prev Cardiol. 2016 Nov;23(16):1715-1733. doi: 10.1177/2047487316657669. Epub 2016 Jun 27. PMID 27353128